CLINICAL TRIAL: NCT04797559
Title: Suprazygomatic Maxillary Nerve (SZMN) Blocks for Pain Control in Pediatric Patients Undergoing T&A: Randomized Controlled Trial ]
Brief Title: SZMN Blocks for Pain Control in Pediatric Patients Undergoing T&A
Acronym: SZMN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Chi-Ho Ban Tsui, Professor, Stanford University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 60450
Record Dates: First submitted 2021-03-10; First posted 2021-03-15 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Postoperative Pain; Opioid Use
Keywords: SZMN Block; Tonsillectomy and Adenoidectomy; Regional Anesthesia
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Patients in the interventional group will receive a total of 5 mL of local anesthetic bilaterally near their temples.
Who Masked: Participant, Care Provider
Masking Description: Both groups will receive a small circular band-aid on their temples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SZMN Treatment Group (Experimental): Patients randomized into the SZMN-treatment group will receive a bilateral single injection SZMN block under general anesthesia in the operating room. The injection will occur through the pterygomaxillary fissure into the pterygomaxillary fossa. Patients will receive 5 ml of local anesthestic per side.
  Interventions: Procedure: SZMN Block
- Control Group (No Intervention): Patients in this group will receive the standard of care for T&A procedures within the pediatric population.

INTERVENTIONS:
Procedure: SZMN Block — Suprazygomatic Maxillary Nerve (SZMN) Blocks bilaterally near the temples of the patient
  Arms: SZMN Treatment Group

SUMMARY:
The suprazygomatic maxillary nerve (SZMN) block is a well-established, safe and effective regional technique for pain management following cleft palate procedures, however, have not been studied for patients undergoing tonsillectomy and adenoidectomy (T&A) procedures. The goals of this study are to determine if SZMN block can be utilized for pain control and decrease morbidity in pediatric patients undergoing T&A.

DETAILED DESCRIPTION:
Patients between 6 months and 18 years undergoing T&A surgical procedures will be reviewed for potential study enrollment. If participants agree to participate, they will be randomized into either the suprazygomatic maxillary nerve (SZMN) block treatment cohort or the control cohort i.e standard of care.

After anesthesia induction, patients randomized into the SZMN- treatment group will receive a bilateral single injection SZMN block under general anesthesia in the operating room. The injection will occur near the temples above the cheek bones.

Participants enrolled into the control group will receive standard of care with no changes to their anesthetic or surgical care. Both groups will be asked for their verbal pain scores in the PACU and we will track their opioid consumption throughout the next few days after their procedure.

ELIGIBILITY:
Inclusion Criteria:

* Ages 0-18
* Give consent/parental consent to participate in study
* Patients undergoing tonsillectomy and adenoidectomy

Exclusion Criteria:

* Participants who do not consent or have parental consent
* Patients who are clinically unstable or require urgent/emergent intervention
* Patients under age 6 months

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2021-11-29 (Actual); Primary Completion 2023-04-19 (Actual); Study Completion 2023-04-19 (Actual)

PRIMARY OUTCOMES:
Post Surgical Pain | 7 days after surgery
  Patients will rate their pain on a 0-10 scale

SECONDARY OUTCOMES:
Opioid Consumption | 1-3 hours after surgery (during the patient's stay in post-anesthesia care unit)
  Pain medications consumed by patients will be collected

CONTACTS AND LOCATIONS:
Overall Officials: Ban C Tsui, MD, Study Director — Professor; Carole Lin, MD, Principal Investigator — Pediatric Anesthesiologist
Locations (1):
- Lucille Packard Children's Hospital, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chiono J, Raux O, Bringuier S, Sola C, Bigorre M, Capdevila X, Dadure C. Bilateral suprazygomatic maxillary nerve block for cleft palate repair in children: a prospective, randomized, double-blind study versus placebo. Anesthesiology. 2014 Jun;120(6):1362-9. doi: 10.1097/ALN.0000000000000171. PMID 24525630
- [Result] Grainger J, Saravanappa N. Local anaesthetic for post-tonsillectomy pain: a systematic review and meta-analysis. Clin Otolaryngol. 2008 Oct;33(5):411-9. doi: 10.1111/j.1749-4486.2008.01815.x. PMID 18983373
- [Derived] Lin C, Abboud S, Zoghbi V, Kasimova K, Thein J, Meister KD, Sidell DR, Balakrishnan K, Tsui BCH. Suprazygomatic Maxillary Nerve Blocks and Opioid Requirements in Pediatric Adenotonsillectomy: A Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2024 Jul 1;150(7):564-571. doi: 10.1001/jamaoto.2024.1011. PMID 38780948